CLINICAL TRIAL: NCT06300788
Title: Inorganic Pyrophosphate Homeostasis (PPi) in Pediatric Chronic Kidney Disease - PPi-DIA
Brief Title: Inorganic Pyrophosphate Homeostasis (PPi) in Pediatric Chronic Kidney Disease
Acronym: PPi-DIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-AOI-02
Record Dates: First submitted 2024-02-13; First posted 2024-03-08 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Pyrophosphate, Fetuin A, IL1, IL6, TNFalpha, Control
Keywords: Pyrophosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CKD group (Experimental): Patient with chronic kidney disease
  Interventions: Other: PPI and T50 dosing
- Dialysis group (Experimental): Dialysis patients (hemodialysis or peritoneal dialysis)
  Interventions: Other: PPI and T50 dosing
- kidney transplant group (Experimental): Kidney transplant patients
  Interventions: Other: PPI and T50 dosing
- Control group (Active Comparator): Control group of patients with normal renal function
  Interventions: Other: PPI and T50 dosing

INTERVENTIONS:
Other: PPI and T50 dosing — Sampling for PPI determination and T50 in blood and urine.

SUMMARY:
The investigator aim to identify the role of inorganic pyrophosphate and other anti-calcifying molecules in vascular disease in children with chronic kidney disease, with a view to developing therapeutic approaches aimed at limiting the onset of vasculopathy.

DETAILED DESCRIPTION:
The study of pro- and anti-calcifying molecules in children with chronic kidney disease will be carried out using dosages made on serum in comparison with the dosage of these same molecules in control children matched according to age and sex. without chronic kidney disease. An evaluation of vascular function by clinical (auscultation, palpation) and ultrasound techniques (measurement of intima-media thickness and measurement of pulse wave velocity) will also be carried out in children with chronic kidney disease and compared to norms of children without chronic kidney disease. These evaluations aim to improve understanding of the pathophysiology of vascular calcification and thus open up therapeutic perspectives in these children.

ELIGIBILITY:
Inclusion Criteria:

All groups :

* Minor patients (<18 years)
* Patients of both sexes
* Informed patients and parents who have signed the informed consent form
* Patients affiliated to social security

Control group :

- Patients with no particular pathology undergoing surgery and receiving a preoperative check-up

CKD groups :

* Patients on dialysis for more than 3 months, regardless of technique
* Kidney transplant patients
* Patients with CKD, whatever the cause

Exclusion Criteria:

* Progressive cancer or kidney disease
* Treatments that may modify PPi concentration (e.g. bisphosphonates)

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2026-11-27 (Estimated); Study Completion 2026-11-27 (Estimated)

PRIMARY OUTCOMES:
Plasma pyrophosphate concentration [PPi]pl in children with CKD | 18 months
  Compare plasma pyrophosphate concentration [PPi]pl between children with CKD (dialysis group and non-dialysis, non-transplant group) and [PPi]pl of children with normal renal function.
  Plasma PPi concentration during fasting sampling; (μmol/L) by a proprietary assay developed at LP2M.
  We will match the 3 MRC groups with their respective control groups according to age, sex and pubertal stage.

SECONDARY OUTCOMES:
Plasma pyrophosphate [PPi]pl concentration in children with renal transplantation | 18 months
  To compare the plasma pyrophosphate [PPi]pl concentration of children with renal transplantation with that of children with dialyzed CKD and children with normal renal function.
  Plasma PPi concentration during fasting sampling; (μmol/L) by a patented assay developed at LP2M.
Markers of phosphocalcic metabolism | 18 months
  To investigate an association between plasma PPi concentration and markers of phosphocalcium metabolism in patients in the 3 MRC groups: dialysis, transplant and non-dialysis/non-transplant).
  The T50 (Serum protection against vascular calcification) marker of phosphocalcium metabolism will be studied.
Urinary PPi concentration | 18 months
  To search for an association between urinary Ppi concentration and markers of phosphocalcium metabolism in patients in the 3 MRC groups: dialysis, transplant and non-dialysis/non-transplant).
  Urinary PPi concentration will be measured by a patented assay developed at LP2M.
Markers of vascular damage in CKD | 18 months
  To look for an association between blood and urine Ppi concentrations and markers of vascular damage in MRC in each of the 3 MRC groups.
  The following markers of vascular damage in CKD will be studied:
  * Measurement of aortic stiffness by ultrasound aortic pulse wave velocity
  * Measurement of carotid intima-media thickness by ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nice - Hôpital de l'Archet 2, Nice, Alpes-Maritimes, France